CLINICAL TRIAL: NCT03158909
Title: Randomized Clinical Trial to Evaluate the Effect of a Non-pharmacological Intervention to Prevent Delirium Among Elderly In-patients
Brief Title: Trial of a Non-pharmacological Intervention to Prevent Delirium Among Elderly In-patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 160529
Record Dates: First submitted 2017-05-11; First posted 2017-05-18 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Delirium
Keywords: Eyemask; Earplugs
MeSH Terms: conditions — Delirium | interventions — Ear Protective Devices; Time

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Patients in this group will receive eyemask and earplugs, for use during the night, and orientations about space and time, every night.
  Interventions: Device: Eyemask and earplugs; Other: Orientation about space and time
- Orientation about space and time (Active Comparator): This group will receive orientations about space and time olny, every night.
  Interventions: Other: Orientation about space and time

INTERVENTIONS:
Device: Eyemask and earplugs — Eyemask and earplugs for use during the night, to improve sleep.
  Arms: Interventional
Other: Orientation about space and time — Information and orientation about space and time, given every night.

SUMMARY:
This study evaluates the effect of earplugs and eyemask for delirium prevention among elderly in-patients. Half of patients will receive earplugs and eyemask for use during the night and information about orientation to time and space every night, while the other half will receive only the time and space orientations.

DETAILED DESCRIPTION:
Delirium is an acute neuropsychiatric syndrome usually associated with a general medical condition. Its prevalence is high among hospitalized elderly patients and is generally underdiagnosed. Delirium is associated with prolonged hospitalization, increased mortality, institutionalization, falls, cognitive and functional decline and also with higher economic costs. The etiology of delirium is multifactorial, including excessive sensorial stimulation and disruption of the sleep-wake cycle as triggering factors.

The aim of this study is evaluate the effect of earplugs and eyemask for delirium prevention among elderly in-patients of a brazilian university hospital. This will be a partially blinded clinical trial, in wich both control and intervention group will receive information about orientation to time and space every evening, and intervention group will also receive earplugs and eyemask for use during the night. The primary outcome will be the occurrence of delirium.

ELIGIBILITY:
Inclusion Criteria:

* In-patients, expected to stay for at least 24 hours.
* Understand and consent in participating in the study and sign the consent form.
* 60 years of age, or older.
* Visual and auditory acuity sufficient to perform cognitive tests.

Exclusion Criteria:

* Diagnosis of delirium in the selection visit.
* Glasgow Coma Scale less than 15 in the selection visit.
* PRISMA-7 ≤3 patient will be excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Incident cases of delirium. | Patients will be followed until diagnosis of delirium, death, discharge from hospital or transfer to another unit, up to 15 days from the inclusion in the study.
  The short version of the Confusion Assessment Method (Short-CAM) will be used.

SECONDARY OUTCOMES:
Sleep quality | Daily as long the patient is still being followed, up to 15 days from the inclusion in the study.
  A questionnaire composed of questions will be used.
Safety of the intervention. | Daily as long the patient is still being followed, up to 15 days from the inclusion in the study.
  Record of adverse effects.
Acceptance, confort and adherence to the intervention. | After every night of eyemask and earplugs use, up to 15 days from the inclusion in the study.
  A four questions questionnaire will be used.
Use of psychotropic drugs. | Patients will be followed until diagnosis of delirium, death, discharge from hospital or transfer to another unit, up to 15 days from the inclusion in the study.
  Record of psychotropic drugs prescribed.
Time of hospital stay. | Until hospital discharge, up to 6 months from inclusion in the study.
  The total time of hospital stay will be recorded.
Evaluation of the sleep-wake cycle. | Daily as long the patient is still being followed, up to 15 days from the inclusion in the study.
  Actigraphy: A technique for assessing the sleep-wake cycle that allows the recording of motor activity through limb movements for 24 hours or more.
Urinary 6-sulfatoxymelatonin levels. | 48 hours after admission (first urine of the day)
  Urinary 6-sulfatoxymelatonin levels 48 hours after admission (first urine of the day).

CONTACTS AND LOCATIONS:
Overall Officials: Artur S Schuh, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil

IPD SHARING:
Plan to Share IPD: Undecided